CLINICAL TRIAL: NCT07404137
Title: A Randomized, Single Dose, Crossover Study to Assess the Effect of Food on the Pharmacokinetics of Single Dose, Orally Administered, Combined Zibotentan/Dapagliflozin in Healthy Participants
Brief Title: A Study to Investigate the Concentrations of Zibotentan and Dapagliflozin in Blood When Given With and Without Food
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D4327C00003
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants
Keywords: Chronic kidney disease; Pharmacokinetics; Food effect; Fixed-dose combination
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment AB (Experimental): Participants will receive single dose of Zibotentan/Dapagliflozin FDC after an overnight fast of at least 10 hours (Treatment A). After a washout period, participants will receive another single dose of Zibotentan/Dapagliflozin FDC 30 minutes after having a high-fat, high-calorie standardized meal (Treatment B).
  Interventions: Drug: Zibotentan/Dapagliflozin FDC
- Treatment BA (Experimental): Participants will receive single dose of Zibotentan/Dapagliflozin FDC 30 minutes after having a high-fat high-calorie standardized meal (Treatment B). After a washout period, participants will receive another single dose of Zibotentan/Dapagliflozin FDC after an overnight fast of at least 10 hours (Treatment A).
  Interventions: Drug: Zibotentan/Dapagliflozin FDC

INTERVENTIONS:
Drug: Zibotentan/Dapagliflozin FDC — Zibotentan/Dapagliflozin FDC will be administered as an oral tablet.

SUMMARY:
The purpose of this study is to investigate the concentrations of zibotentan and dapagliflozin in blood when given with and without food in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomized, 2-period, 2-treatment, crossover study in healthy participants.

This study will measure the impact of food on the pharmacokinetics (PK) of combined zibotentan/dapagliflozin for the to be marketed fixed-dose combination (FDC) formulation (study intervention).

The study will comprise of, (i) A screening period (ii) 2 treatment periods (iii) A final follow-up visit.

All participants will receive a single dose of the study intervention once under fasted condition (Treatment A) and once under fed condition (Treatment B).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-childbearing potential. Participants with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg (inclusive) at Screening.

Exclusion Criteria:

* History of any clinically important disease or disorder.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma.
* Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results or other laboratory values or vital signs.
* Any positive result on screening for serum Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis C virus (HCV) antibody, or Human immunodeficiency virus (HIV) (Type 1 and 2) antibodies.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* History or ongoing allergy/hypersensitivity, to Sodium-Glucose Cotransporter-2 Inhibitors (SGLT2i- eg, dapagliflozin, empagliflozin), or zibotentan or other Endothelin Receptor Antagonist (ERAs- eg, ambrisentan, atrasentan,bosentan), or any of the excipients in the zibotentan/dapagliflozin tablets.
* Participants who have previously received zibotentan.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) | At predefined intervals from Day 1 to Day 4 for both treatment periods
  To investigate the effect of a high fat, high calorie meal, in comparison to fasting conditions, on the PK of zibotentan/dapagliflozin FDC after a single oral dose in healthy participants.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | At predefined intervals from Day 1 to Day 4 for both treatment periods
  To investigate the effect of a high fat, high calorie meal, in comparison to fasting conditions, on the PK of zibotentan/dapagliflozin FDC after a single oral dose in healthy participants.
Maximum observed drug concentration (Cmax) | At predefined intervals from Day 1 to Day 4 for both treatment periods
  To investigate the effect of a high fat, high calorie meal, in comparison to fasting conditions, on the PK of zibotentan/dapagliflozin FDC after a single oral dose in healthy participants.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to end of study visit, for a total of approximately 5 weeks
  To further assess the safety and tolerability of single doses of zibotentan/dapagliflozin FDC in healthy participants.
Apparent total body clearance (CL/F) | At predefined intervals from Day 1 to Day 4 for both treatment periods
  To further evaluate the PK of zibotentan/dapagliflozin FDC after a single oral dose in healthy participants.
Apparent volume of distribution based on the terminal phase (Vz/F) | At predefined intervals from Day 1 to Day 4 for both treatment periods
  To further evaluate the PK of zibotentan/dapagliflozin FDC after a single oral dose in healthy participants.
Time to reach maximum observed concentration (tmax) | At predefined intervals from Day 1 to Day 4 for both treatment periods
  To further evaluate the PK of zibotentan/dapagliflozin FDC after a single oral dose in healthy participants.
Terminal elimination half-life (t½λz) | At predefined intervals from Day 1 to Day 4 for both treatment periods
  To further evaluate the PK of zibotentan/dapagliflozin FDC after a single oral dose in healthy participants.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/